CLINICAL TRIAL: NCT05807152
Title: Furosemide-induced Diuresis With Matched Dehydration Compared to Standard Diuretic Therapy in Acute Heart Failure and Overt Fluid Overload
Brief Title: Furosemide-induced Diuresis With Matched Dehydration Compared to Standard Diuretic Therapy in Patients With Acute Heart Failure and Overt Fluid Overload
Acronym: MYTHOS-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Piergiuseppe Agostoni, Professor, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCM 964
Record Dates: First submitted 2023-02-21; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Acute Decompensated Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Furosemide infusion (standard treatment)
- RenalGuard group (Experimental): Furosemide infusion with matched de-hydration
  Interventions: Device: RenalGuard device

INTERVENTIONS:
Device: RenalGuard device — Patients will be given an intravenous loading dose of 40 mg of furosemide and continuous infusion of furosemide based on baseline eGFR. An additional bolus of 40 mg of furosemide will be administered and the infusion rate increased according to the same protocol of the control group (Figure 1). The venous peripheral cannula will be connected with the extracorporeal circuit of the RenalGuard System (PLC Medical Systems Inc., MA) for fluid infusion. The RenalGuard System is capable of delivering sterile replacement solution to a patient in an amount matched, or higher or lower, to the volume of urine produced by the patient. Thus, in the RenalGuard group, estimated daily targeted negative fluid balance will be utilized to define, for each patient, hourly negative fluid balance to be set in the RenalGuard system display.
  Arms: RenalGuard group

SUMMARY:
Acute decompensated heart failure (ADHF) is a complex clinical syndrome caused by cardiac abnormalities compromising the ability of the heart to provide a blood supply adequate to the metabolic needs of peripheral tissues. ADHF is characterized by systemic and pulmonary fluid retention, with weight gain, peripheral edema, needing diuretic therapy. Moreover, ADHF is associated with neurohormonal hyper-activation with enhanced sympathetic nervous and renin-angiotensin-aldosterone systems stimulation, that sustain the vicious circle of cardiac dysfunction and fluid retention.

The administration of high doses of diuretics, usually required in ADHF treatment, can induce hypovolemia-induced neurohormonal activation and transient deterioration of kidney function, that, in turn, counteracts the effect of diuretics and limits recovery from fluid overload.

The investigators hypothesized that, in patients with ADHF, a more controlled and physiologically-oriented dehydration may blunt diuretic-associated neurohormonal activation, thus providing a safer and more sustained clinical benefit. This controlled dehydration can be achieved by combining furosemide with the RenalGuard System (see The RenalGuard™ System Operator's Manual for specific instructions in setting up and running the device). To date, no data have been provided regarding the potential beneficial effect of this therapeutic strategy in patients with ADHF and fluid overload. Much of the evidences on the use of the RenalGuard system comes from the clinical setting of acute kidney injury (AKI) prevention in patients undergoing intravascular contrast exposure. In this specific field, furosemide-induced high-volume diuresis with concurrent maintenance of intravascular volume through matched hydration, by the RenalGuard System, is now considered by current Guidelines a recommended strategy for AKI prevention in patients with chronic renal failure undergoing coronary interventional procedures. Based on this experience, the investigators will assess the safety and efficacy of this known system capable of delivering intravenous fluid in an amount exactly pre-determined, considering the volume of urine produced by the patient and precisely weighed by the system. This could prevent hypovolemia that may occur in response to high-volume diuresis induced by furosemide. The researchers will perform a spontaneous, prospective, randomized trial aiming at investigating the effect of combined furosemide-induced diuresis and automated matched dehydration, compared with standard furosemide administration in ADHF patients with fluid overload.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* New York Heart Association (NYHA) functional class III or IV
* estimated weight gain due to peripheral fluid overload >4 kg
* admission BNP values >400 pg/ml if in sinus rhythm and >600 pg/ml if in atrial fibrillation

Exclusion Criteria:

* inability to provide informed consent
* acute pulmonary edema, cardiogenic shock
* end-stage renal disease (Stage V) or need for renal replacement therapy
* ongoing treatment with Entresto (BNP not reliable)
* need for inotropic/vasopressor drug support
* contraindications to placement of a Foley catheter.
* Known hypersensitivity to furosemide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Daily serum creatinine measurement during study treatment for assessment of acute kidney injury occurrence | Daily, up to 72 hours
  Blood sample for creatinine evaluation will be performed daily

SECONDARY OUTCOMES:
Daily weight decrease during study treatment | Daily, up to 72 hours
  Weight evaluation will be performed daily

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Irccs, Milan, Italy